CLINICAL TRIAL: NCT03740399
Title: Effect of Modified 45-degree Head-up Tilt Position in Cesarean Operation to the Success of Spinal Anesthesia
Acronym: cesarean
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sevtap Hekimoglu Sahin, Clinical Professor, Trakya University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TÜTF-BAEK 2018/79
Record Dates: First submitted 2018-10-19; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Regional Anesthesia Morbidity
Keywords: sitting position; lateral decubitus position; spinal block
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group sitting (Active Comparator): we are performing spinal anesthesia in sitting position pregnant patients
  Interventions: Procedure: spinal anesthesia
- Group lateral decubitus position (Active Comparator): we are performing spinal anesthesia in lateral decubitus position pregnant patients
  Interventions: Procedure: spinal anesthesia
- Group Modified 45-degree head-up tilt (Active Comparator): we are performing spinal anesthesia in Modified 45-degree head-up tilt position pregnant patients
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — Investigators will perform spinal anesthesia for section

SUMMARY:
The success of the application of spinal block in 3 different application as the sitting position, side decubitus position and 45 degrees head upside side decubitus position will be evaluated.

DETAILED DESCRIPTION:
180 patients in ASA I-II risk group between the ages of 18-50 will be included in the study.The success of the application of spinal block in 3 different application as the sitting position, side decubitus position and 45 degrees head upside side decubitus position will be evaluated. Anatomical features of height, weight, block application of the patients will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* caesarean section
* 18-50 years old
* ASA I-II risk

Exclusion Criteria:

* heart failure
* patient's refusal
* thrombocytopenia
* coagulation disorder
* heart valve diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant womans
Enrollment: 180 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-03-28 (Estimated); Study Completion 2019-06-28 (Estimated)

PRIMARY OUTCOMES:
spinal anesthesia success | spinal anesthesia success will be 15 minutes in intraoperative
  The free flow of clear cerebrospinal fluid (CSF) upon first attempt was considered to be evidence of a successful LP.

CONTACTS AND LOCATIONS:
Overall Officials: Sevtap Hekimoglu Sahin, Proffesor, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Centrum, Turkey (Türkiye)